CLINICAL TRIAL: NCT03672955
Title: Advanced Ultrasound Methods in the Assessment of Carotid Plaque Instability.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Mona Skjelland, Consultant, Associate professor, Oslo University Hospital
Other Study IDs: 2014/1468
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Internal Carotid Artery Stenosis With Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Carotid artery plaques removed by treatment with carotid endarterectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this project is to assess if advanced ultrasound methods such as SMI (Superb microvascular Imaging) and SWE (Shear Wave Elastography) can identify intraplaque neovascularization and plaque tissue stiffness in carotid artery plaques and relate these results to ipsilateral cerebrovascular symptoms.

The secondary aim of this project is to assess the level of agreement between the structural plaque characteristics assessed by advanced ultrasound examinations such as SMI, SWE, CEUS (Contrast enhanced ultrasound), GSM (Plaque gray-scale-median) and carotid MRI, metabolic activity of plaque assessed by 18F-FDG PET/CT with histology as the gold standard. Findings from the methods mentioned above will be related to cerebrovascular symptoms, blood tests (cholesterol-tot, LDL, HDL, CRP, leukocytes, glucose, HbA1c) and other cardiovascular risk factors at inclusion and upon 1 year follow up.

DETAILED DESCRIPTION:
The project will include 3 studies:

Study 1:

Analyse the correlation between SMI assessed neovascularization and degree of stenosis in symptomatic patients with high-grade (>50%) carotid stenosis versus asymptomatic patients with high-grade (>50%) carotid stenosis.

All patients upon inclusion will undergo:

* Clinical, neurological evaluation
* Blood tests
* SMI, CEUS and SWE ultrasound
* Carotid MRI
* PET (subgroup)
* DW-MRI
* Histological assessments after the removal of plaque at carotid endarterectomy (CEA).

Study 2:

SMI and vascular events. Asymptomatic patient's follow-up at 12 months:

* Clinical neurological evaluation
* Blood test
* SMI, CEUS, SWE ultrasound
* Carotid MRI
* PET (subgroup)

Study 3:

This study will use the same patient pool described in study 1 undergoing the previously described procedural examinations upon inclusion and at one year follow up. Quantification of stiffness/elasticity in the artery wall will be performed and compared to plaque echogenicity measured as GSM . These results will be correlated to histology of the carotid plaque after trombendarterectomy, risk markers in blood (lipids, HbA1c, CRP, leukocytes), other cardiovascular risk markers (hypertension, diabetes, nicotine) and cerebrovascular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerotic carotid stenosis >50% with or without cerebrovascular symptoms.

Exclusion Criteria:

* Malignancies
* Inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • All patients with an atherosclerotic carotid stenosis >50% admitting department of neurology, Oslo University Hospital, Rikshospitalet as an in-patient or an out-patient will be considered for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Raised neovascularization and increased stiffness of the carotid artery wall are correlated to cerebrovascular symptoms and raised level of some plasma markers. | one year
  Ultrasound (including SMI, CEUS, SWI), blood test, clinical symptoms and cerebral MRI at inclusion and at one year follow-up

SECONDARY OUTCOMES:
Increased neovascularization in the carotid artery wall assessed by SMI ultrasound is correlated to cerebrovascular symptoms, ischemic lesions on cerebral MR, increased level of some plasma markers and increased vascularization on carotid plaques | At inclusion
  Ultrasound, blood tests, clinical assessment, cerebral MRI, histology of carotid artery plaques (if treated with carotid endarterectomy)
Increased neovascularization in the carotid artery wall assessed by SMI ultrasound is correlated to cerebrovascular symptoms, ischemic lesions on cerebral MR and increased level of some plasma markers at one year follow-up | 1 year
  Clinical assessment, ultrasound, cerebral MRI, blood tests, histology if removed carotid plaque
Increased stiffness in the carotid artery wall assessed by ultrasound (GSM) is correlated to cerebrovascular symptoms and increased level of some plasma markers at one year follow-up | 1
  Clinical assessment, ultrasound, cerebral MRI, blood tests, histology if removed carotid plaque

CONTACTS AND LOCATIONS:
Overall Officials: Mona Skjelland, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway